CLINICAL TRIAL: NCT07157358
Title: Online Medical Hypnosis Exercises to Improve Mental Health in Primary School Children and Prevent Future Mental Health Issues
Acronym: Breinbaas
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Collaborators: Leiden University (Other)
Responsible Party: Principal Investigator, Arine Vlieger, Pediatrician, MD, PhD, St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NL 87558.100.24
Record Dates: First submitted 2025-08-22; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Healty Volunteers
Keywords: mental health; primary school; hypnosis; self-esteem; resilience
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled open-label study with a duration of six months. Children will be randomized to start immediately with the online program with hypnosis exercises o iprove mental well being (Group A) or after 6 months (group B). Group B will therefore be the control group of A.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Childnre in group A will listen daily for 6 weeks to different hypnosis recordings aiming at the increase of self-esteem, resilience, and mental health in general.
  Interventions: Behavioral: standardized audio hypnosis recordings for healthy children at primary school
- Group B (No Intervention): These children will start listening to the exercises after 6 months, which is already the end of the study. Therefor, their scores in the first 6 months are the controls to group A.

INTERVENTIONS:
Behavioral: standardized audio hypnosis recordings for healthy children at primary school — 8 different audio hypnosis recordings hat chidlren will listen too at a daily basis (one recording per day)
  Arms: Group A

SUMMARY:
The goal of this trial is to learn if listening daily to online hypnosis exercises helps to improve mental health and self-esteem in primary school children. In the future we also hope to see if it can prevent feelings of depession or anxiety when these children have become teenagers.

The main questions it aims to answer are:

1. can daily listening to these exercsies improve self-esteem, resilience and mental health of children 10-11 years compared to children who do not listen to these exercises?
2. can listening to these exercsies prevent future metal health problems like feelings of depression or anxiety.

Researchers will compare a group of children (10-11 years) who will listen daily to the exercises for 2 months with a group who will do that 6 months later.

Participants will:

Listen daily to a hypnosis exercise of maximum 15 minutes. Fill out questionnaires on self-esteem, resilience and mental health before during and after the study.

DETAILED DESCRIPTION:
SUMMARY

Rationale:

Early adolescence marks a crucial period for the development and onset of mental health problems, which often manifest as disorders in the course of adulthood if they are not dealt with early on. Moreover, there is an increased prevalence of disorders like anxiety and depression in adolescence. Prevention of these mental health problems is of great importance.

Objective: The primary objective is to study the effect of daily listening for 6 weeks to the Breinbaas hypnosis recordings on selfesteem compared to controls. Secondary objective(s) are studying the effect of daily listening to the Breinbaas hypnosis recordings for 6 weeks on change in resilience, psychosocial functioning, overall stress level, and other effects like sleep compared to controls. Study design: This is a randomized controlled open-label study with a duration of six months. Children will be randomized to start immediately with the online program (Group A) or after 6 months (group B). Group B will therefore be the control group of A.

Study population: Children from grade 6 or 7 of the participating primary schools will be invited to participate. Schools will be recruited in 3 areas in the Netherlands.

Intervention: The online Breinbaas academy program consists of hypnosis audio recordings that children will listen to on every schoolday for six weeks. The hypnosis audio recordings aim to improve children's mental health.

Main study parameters/endpoints: Children fill out questionnaires at baseline, 6 weeks and 6 months about the child's self-esteem, psychosocial functioning, resilience, stress levels, and sleep.

ELIGIBILITY:
Inclusion Criteria: In order to be eligible to participate in this study, a subject must meet all of the following criteria:

1. Fluent in Dutch
2. Attending group 6 or 7 of a regular primary school in the Netherlands
3. Permission of the parents to listen daily to one of the Breinbaas hypnosis exercises (maximum 20 minutes per day)
4. Access to an electronic device to listen to the Breinbaas exercises (phone, tablet, computer) -

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

1. Children treated with hypnotherapy in the three years preceding potential inclusion
2. Children currently receiving psychological treatment

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 345 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Difference in change in self-esteem between group A and B. | difference between baseline and the end of listening to the exercises at 6 weeks.
  The primary objective is to study the effect of daily listening for 6 weeks to the hypnosis recordings on the change in self-esteem compared to controls 6 weeks after baseline. It will be measured by the Rosenberg Self Esteem scale for Children. This gives a score between 0 to 30 and higher scores mean more self-esteem.

SECONDARY OUTCOMES:
Improvement in resilience on short and long term. | CD-RISC will measured between baseline and six weeks and between baseline and after 6 months.
  Difference in improvement in resilience as measured by the Connor-Davidson Resilience Scale for Children (CD-RISC) between group A and Group B. The Connor-Davidson Resilience scale (CD-RISC) comprises of 25 items, each rated on a 5-point scale (0-4), with higher scores reflecting greater resilience.
Improvement in psychosocial functioning on short and long term.. | The difference in SDQ will be measured between baseline and six weeks, and between baseline and after 6 months.
  Change in improvement in psychosocial functioning as measured by the Strength and Difficulties Questionnaire (SDQ) between group A and B. The SDQ asks about 25 attributes, some positive and others negative. These 25 items are divided between 5 scales:
  1. emotional symptoms (5 items)
  2. conduct problems (5 items)
  3. hyperactivity/inattention (5 items)
  4. peer relationship problems (5 items)
  5. prosocial behaviour (5 items) All questions result in 1 to 4 points with higher scores reflecting more problems.
Stress reduction at short and long term. | The CSQ-CA will be measured at baseline, 6 weeks, and 6 months in both groups.
  Change in stress will be compared between group A and B. They are measured by the Chronic Stress Questionnaire for children and adolescents (CSQ-CA) (Stress Vragenlijst Voor Kinderen). It consists of 19 items, including "I often overthink things" and "Ifeel like I have to do too many things at the same time". The items have to be scored on a 4-point scale from "this does not apply to me at all", "this usually does not apply to me", thus usually applies to me", to "this completely applies to me". Higher scores reflect more stress.

OTHER OUTCOMES:
Side-effects of listening to hypnosis exercises | This will be measured at T = 6 weeks.
  Children will be asked if they had noticed any side-effects of using the program. Also, the number of times a child contacts the study team for side effects will be noted.
Treatment adherence | This will be monitored during the phase that the chidlren are listening, which is 6 weeks.
  The app, providing the hypnosis exercises, will monitor how often the children have listened to one of the exercises. Good treatment adherence will be defined as listening at least 4 times a week during 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Arine M Vlieger, MD,PhD, Principal Investigator — St. Antonius Hospital
Locations (1):
- University Leiden, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be shared

REFERENCES:
- [Background] Rutten JMTM, Vlieger AM, Frankenhuis C, George EK, Groeneweg M, Norbruis OF, Tjon A Ten W, van Wering HM, Dijkgraaf MGW, Merkus MP, Benninga MA. Home-Based Hypnotherapy Self-exercises vs Individual Hypnotherapy With a Therapist for Treatment of Pediatric Irritable Bowel Syndrome, Functional Abdominal Pain, or Functional Abdominal Pain Syndrome: A Randomized Clinical Trial. JAMA Pediatr. 2017 May 1;171(5):470-477. doi: 10.1001/jamapediatrics.2017.0091. PMID 28346581
- See also: This Dutch website gives information on the hypnosis exercises used in this study — https://breinbaasacademy.nl/